CLINICAL TRIAL: NCT00470041
Title: Bioavailability Study of a New Pediatric Formulation of Zidovudine/Lamivudine in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Prof. Dr. Luc Van Bortel, University Ghent
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/155
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Lamivudine; Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: administration of two anti-viral drugs (lamivudine and zidovudine) from a new oral formulation

SUMMARY:
Description: To investigate bioavailability of two anti-viral drugs (lamivudine and zidovudine) from a new oral formulation (trial formulation) especially designed for pediatric use.

Interventions: 12 healthy volunteers will receive in a cross-over design two formulations i.e. the commercially available tablet formulation and the trial formulation. Blood samples (13 over 24 h) will be taken in order to determine the pharmacokinetic profile of the drugs from both formulations and will be compared.

Duration of intervention: 2 days + 7 days of wash-out between both oral administrations.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 55 years, extremes included. Males and females.
* Smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day (or non-smoking) for at least 3 months prior to selection.
* Normal weight as defined by a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is competent and willing to sign informed consent form after being given all the detailed information about the study. Informed consent form signed voluntarily.
* Healthy on the basis of a pre-trial physical examination, medical history, electrocardiogram and the results of blood biochemistry and haematology tests and a urinalysis carried out less than 3 weeks before the first dose.

Exclusion Criteria:

* Subjects presenting anaemia, neutropenia or platelets deficits
* Subjects with kidney failure or renal dysfunction
* Pregnant, lactating females
* History of allergy or hypersensitivity to Zidovudine or Lamivudine.
* History of clinically cardiovascular disease or liver disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
bioavailability of two anti-viral drugs (lamivudine and zidovudine) from a new oral formulation (trial formulation) especially designed for pediatric use | over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Luc Van Bortel, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be